CLINICAL TRIAL: NCT04513132
Title: A Study on Targeted Intervention for Insight in Patients with First Episode and Clinical High Risk of Schizophrenia Based on Theta Oscillation in Anterior Cingulate Cortex
Brief Title: Targeted Intervention Study of DTMS on Impaired Insight in Early Psychosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because this research is a modification of a previous study that was not obtained, and the intervention method has changed significantly, we are considering withdrawing this study and reapplying.
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DTMS2024
Record Dates: First submitted 2020-08-05; First posted 2020-08-14 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2023-01

CONDITIONS: Impaired Insight
Keywords: Insight; Deep transcranial magnetic stimulation; Self monitoring; Anterior cingulate cortex; Middle temporal gyrus; Theta oscillation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to different montage of stimulation, including deep transcranial magnetic stimulation (active-dTMS) and sham stimulation (sham-dTMS).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are blind to the dTMS montage. Researchers in this study will include clinical evaluators, laboratory inspectors, dTMS operators, and statistical analysis. Before unblinding, each group of researchers will have no access to the information collected by the other groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- active-CHR (Active Comparator): Participants will be intervened with deep transcranial magnetic stimulation (dTMS).
  Interventions: Device: active-dTMS
- sham-CHR (Sham Comparator): Participants, as a control group, will receive sham stimulation.
  Interventions: Device: sham-dTMS
- active-FES (Active Comparator): Patients with first-episode schizophrenia will be intervened with deep transcranial magnetic stimulation (dTMS).
  Interventions: Device: active-dTMS
- sham-FES (Sham Comparator): Patients with first-episode schizophrenia, as a control group, will receive sham stimulation.
  Interventions: Device: sham-dTMS

INTERVENTIONS:
Device: active-dTMS — The dTMS using H-coil with 5Hz stimulate ACC. The sessions of dTMS will be conducted twice daily for 5 consecutive days, and twice sessions of a day will be separated by 3 hours at least.
  Arms: active-CHR; active-FES
Device: sham-dTMS — The sham-dTMS has the same appearance with the real stimulation coil, which can not generate magnetic field. A sound generator is built in the coil beat to simulate the sound of the real stimulation.
  Arms: sham-CHR; sham-FES

SUMMARY:
Impaired insight is a key factor in the conversion of high-risk individuals to schizophrenia, but there is a lack of targeted interventions. We found that an electroencephalogram (EEG) signal reflecting the function of self monitoring was a potential objective marker of impaired insight. And further functional magnetic resonance imaging (fMRI) analysis showed that the functional connectivity between anterior cingulate gyrus (ACC) and medial temporal gyrus (MTG) was related to insight. Studies have shown that ACC theta oscillation is the key to self monitoring, and theta-alpha phase synchronization between frontotemporal is closely related to cognition. Therefore, this project hypothesized that targeted regulation of ACC theta oscillations could promote theta-alpha phase synchronization and functional connectivity between ACC and MTG, thereby improving patients' insight. The first-episode and high-risk subjects were recruited to detect the theta oscillation of ACC, theta-Alpha phase synchronization and functional connectivity between ACC and MTG using EEG-fMRI. Deep transcranial magnetic stimulation was introduced to regulate ACC theta oscillations. The high-risk subjects were followed up for two years. It was estimated that the theta-alpha phase synchronization of ACC-MTG and insight in the active-dTMS group were significantly improved. And the outcome of the high-risk subjects is better. The project develops neuroregulatory techniques for impaired insight of schizophrenia and is expected to provide a solution for this clinical pain point.

DETAILED DESCRIPTION:
The study will conduct randomized and controlled experimental design, including deep transcranial magnetic stimulation (dTMS) and sham stimulation (SH-dTMS). Each included participant will be given informed consent and then randomly assigned to different montage of stimulation. Participants are blind to the dTMS montage. Researchers in this study will include clinical evaluators, laboratory inspectors, dTMS operators, and statistical analysts. Before unblinding, each group of researchers will have no access to the information collected by the other groups. For example, except the dTMS operators, no one knows which stimulus montage any of the participants receive. The sessions of dTMS will be conducted twice daily for 5 consecutive days, and twice sessions of a day will be separated by 3 hours at least. Clinical assessments and laboratory tests will be administered at baseline and at the end of the last session. After the post-intervention tests, first stage unblinding will be conducted. At this moment, dTMS operators will provide the groups of A and B, but no corresponding montage, to the statistical analysts. After analyzing the differences between the two groups, second stage unblinding will be performed and the results of the clinical trial will be further analyzed by revealing the corresponding stimulus montage of each group. This study will be implemented at a single center, the Shanghai Mental Health Center (SMHC).

ELIGIBILITY:
Inclusion Criteria:

* 14~35 years old;
* Meet the criteria of clinical high risk for psychosis or meet the DSM-V diagnostic criteria for schizophrenia;
* Meeting the following definition of impaired insight;
* Having completed at least six years of primary education;
* Being able to give informed consent, oral or written. Patients under 18 years old give oral consent and their next of kin or legal guardians give written consent.

Exclusion Criteria:

* Participating in any other clinical intervention research;
* Meeting the diagnostic criteria of psychotic disorders (including affective disorders);
* Threshold symptoms are induced by other mental disorders or psychoactive substances;
* Undergoing anti-psychotic medication for more than 2 weeks;
* Being diagnosed as organic brain diseases, or severe somatic diseases;
* Had Experienced traumatic brain injury, and got scores of 7;
* Dementia, or mental retardation (IQ<70);
* Being a condition of scalp infection;
* A pacemaker or other metal implants in the body, pregnancy, or claustrophobia.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in clinical insight | Baseline and immediately after the intervention
  Clinical insight will be assessed using SAI. SAI is a semi-structured interview tools including seven items, with a total score of 14, 0-6 for recognition of illness, 0-4 for relabeling of psychotic phenomena, and 0-4 for treatment compliance. Patients, with less than 3 scores on recognition of illness, 2 on relabeling of psychotic phenomena, and 2 on treatment compliance, are considered to be improved on insight.
Change in error-related negativity | Baseline and immediately after the intervention
  The error-related negativity (ERN) is observed over frontocentral sites within 100 ms following an error response in behavioral tasks, reflecting error-detecting activity, and a reduced ERN indicates reduced error monitoring. EEG epochs were marked with artifacts and excluded from the following ERN analysis if on any electrode, (i) the maximal peak-to-peak amplitude exceeded 100 μV within any moving window (width: 200 ms; step: 50 ms) or (ii) the absolute amplitude exceeded 100 μV at any time point. The calculation for the ERN was based on no fewer than five available epochs with erroneous responses.
Change in Resting-state functional brain connectivity between anterior cingulate cortex (ACC) and middle temporal gyrus (MTG) | Baseline and immediately after the intervention
  Imaging data will be collected on a 3-T Siemens Magnetom Verio syngo MR B17 scanner and a 32-channel head coil, including structural phase and resting stage detection, which will be used to analyze the functional connection between ACC and MTG.

SECONDARY OUTCOMES:
Change in psychopathological symptoms | Baseline and immediately after the intervention
  This study will also observe the psychopathological symptoms, including positive, negative and general symptoms, using PANSS.The reductive ratio of PANSS points will be calculated after dTMS treatment.
Covariant change of clinical insight and psychopathological symptoms | Baseline and immediately after the intervention
  Clinical insight will be assessed using SAI, and the psychopathological symptoms will be measured using PANSS. The correlation of psychopathological symptoms with clinical insight will be analyzed, especially possible covariant change after dTMS treatment.
Change in reality monitoring ability | Baseline and immediately after the intervention
  Reality monitoring ability refers to distinguish internally self-generated information from externally-derived information. The test will be carried out by the experimental paradigm of reality monitoring ability.The stimulus materials are easy to be accepted and understood by patients with mental illness.The material consisted of 48 pairs of familiar pictures and was divided into two tests, each consisting of a learning and a testing phase. In the learning phase, 24 pictures will be presented with different combinations of conditions (four combinations of "perceptive/imaginative × left/right" conditions). In the testing phase, one object will be presented and the participants will be asked to decide whether the other paired object is perceptive or imaginative, or whether the image is positioned on the left or right side of the screen.
Change in theta oscillation in ACC and theta-alpha phase synchronization between ACC and MTG | Baseline and immediately after the intervention
  Theta oscillation and theta-alpha phase synchronization will be recorded using using a magnetic resonance compatible 64 electrode cap (BrainAMP MR, Brain Products, Munich, Germany) based on the international society for electroencephala 10/20 standard system.
Convertion rate of transition into psychosis | 2 year
  This study will use SIPS to identify individuals with CHR and assess the participants' clinical outcomes, including transition into psychosis, symptomatic, remission, and other disorders

CONTACTS AND LOCATIONS:
Overall Officials: Jijun Wang, Doctoral, Study Chair — Shanghai Mental Health Center; Tianhong Zhang, Doctoral, Study Director — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No